CLINICAL TRIAL: NCT05173519
Title: A Prospective, Randomized, Single-blinded Study to Assess the Incidence of Wound Complications Following Total Knee and Hip Arthroplasty in Patients Treated With Two Different Types of Topical Skin Adhesive
Brief Title: Omnibond vs Dermabond
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporarily halted
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Omnibond001
Record Dates: First submitted 2021-11-29; First posted 2021-12-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Omnibond topical skin adhesive (Active Comparator)
  Interventions: Device: Omnibond Topical Skin Adhesive
- Dermabond topical skin adhesive (Active Comparator)
  Interventions: Device: Dermabond Advanced Topical Skin Adhesive

INTERVENTIONS:
Device: Omnibond Topical Skin Adhesive — Application of Omnibond topical skin adhesive to close incision following surgery
  Arms: Omnibond topical skin adhesive
Device: Dermabond Advanced Topical Skin Adhesive — Application of Dermabond topical skin adhesive to close incision following surgery
  Arms: Dermabond topical skin adhesive

SUMMARY:
This prospective, randomized, controlled, blinded clinical trial is designed to assess the incidence of all time and all types of wound-related complications following total joint arthroplasty (TJA) when two different types of topical skin adhesives are used to close the incision.

DETAILED DESCRIPTION:
The aim of this study is to assess the incidence of incision healing complications in patients undergoing primary total knee replacement and total hip replacement treated with either Omnibond or Dermabond advanced topical skin adhesive. All patients undergoing a primary, elective TKA and THA at participating centers that sign a consent form will be followed up for a period of up to 30 days to determine if there are any incision healing complications.

Secondary outcomes will include dry time of the topical skin adhesive, user satisfaction, patient satisfaction, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old
2. Male or non-pregnant, non-lactating, postmenopausal or surgically sterilized females
3. Subjects scheduled to undergo primary, elective total knee arthroplasty or total hip arthroplasty
4. Subjects provide informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information
5. Subjects deemed able to understand and comply with study visit schedule and procedures

Exclusion Criteria:

1. Local skin conditions such as dermatitis, eczema, psoriasis that, in the opinion of the investigator, will make it difficult to assess wound complications or local skin reactions following surgery
2. Pregnant, lactating females, or females of childbearing potential not willing to practice an effective method of contraception
3. Active or previous infection in the skin or the knee or hip to be operated, evidence of gangrene
4. Subjects who have participated in this trial previously and who were withdrawn
5. Subjects with known allergies to product components including cyanoacrylate, formaldehyde, benzalkonium chloride or have known allergies or skin sensitivity to the Convatec Aquacel dressing.
6. Inability or refusal to provide informed consent or follow study and wound care instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
All time wound complications | From surgery to 30 days post-op
  any occurrence of a wound-related complication following surgery

SECONDARY OUTCOMES:
Dry time | From time of initial product placement on the skin to when the entire application is dry to the touch with a gloved hand
  Time to dry (in seconds) between Omnibond vs Dermabond will be collected
User satisfaction with study treatment | Up to 1 hour after study product application
  Visual Analog Scale (VAS) will be used to ask users how satisfied they were with the product. The scale minimum value is 0 and maximum value is 100. The higher the score, the higher the user satisfaction with the study product
Subject satisfaction with study treatment | Up to 14 days following surgery
  Subjects will be asked at the time of first post-operative visit how satisfied they are with their study treatment using a Visual Analog Scale (VAS). The scale minimum value is 0 and maximum value is 100. The higher the score, the higher the patient satisfaction with the study product

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Morrison, MS, Study Director — Center for Innovation and Research Organization
Locations (4):
- United States (4):
  - Columbia University, New York, New York
  - JIS Orthopaedics, New Albany, Ohio
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island